CLINICAL TRIAL: NCT06300372
Title: Ultrasonography-Guided Bilateral Modified Thoracoabdominal Nerve Plane Block With Perichondrial Approach (M-TAPA) For Postoperative Pain Management In Living Liver Donors: Randomized Controlled Study.
Brief Title: Modified Thoracoabdominal Nerve Plane Block In Living Liver Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 2
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Liver Failure; Acute Postoperative Pain
Keywords: Modified Thoracoabdominal Nerve Plane Block; Liver Transplantation; Acute Postoperative Pain
MeSH Terms: conditions — Liver Failure; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Fifty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II, scheduled for living liver donation surgery for liver transplantation will be included in the study. Patients will be randomly divided into two groups (Group A=M-TAPA block group, Group B = control group) including 25 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor and participants will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A=M-TAPA block group (Experimental): M-TAPA plane block will be performed and standard postoperative pain management protocols will be applied.
  Interventions: Procedure: M-TAPA plane block; Procedure: Postoperative pain management
- Group B = control group (Active Comparator): Only standard postoperative pain management protocols will be applied. No plane blocks will be applied
  Interventions: Procedure: Postoperative pain management

INTERVENTIONS:
Procedure: M-TAPA plane block — As the patient is in the supine position, the high-frequency linear US probe (11-12 MHz, Vivid Q) and a 22-G 80-mm needle (Pajunk Sonoplex Nanoline Stim Cannula, Germany) will be placed in a sagittal position at the costochondral junction at the level of the 9th and 10th ribs. After the rib and the external oblique, internal oblique, and transversus abdominis muscles are visualized on USG, using an in-plane technique, the block needle will be advanced and the block location will be confirmed by injecting 5 ml of saline between the internal oblique and transversus abdominis muscles. Once the block location is confirmed, 30 ml of 0.25% bupivacaine (Buvicaine ®) will be applied bilaterally (60 ml in total).
  Arms: Group A=M-TAPA block group
Procedure: Postoperative pain management — For preemptive analgesia, morphine (Morfin ®) 0.05mg/kg and Ibuprofen 400mg IV (Ibuprofen®) will be administered to all patients before the surgical incision. An additional dose of ibuprofen 400mg IV, meperidine (Aldolan ®), and tramadol (Contramal®) 1mg/kg IV will be administered to all patients 30 minutes before wound closure.10 mcg/ml fentanyl containing PCA will be connected to all patients without infusion and boluses 0,35 mcg/kg,15-minute lockout period, maximum 100 mcg per hour. Postoperative patient evaluation will be performed by another anesthesiologist. If the NRS score is ≥ 4, 0.5 mg/kg IV meperidine (Aldolan®)will be administered as a rescue analgesic.

SUMMARY:
Ultrasound-guided Modified Thoracoabdominal Nerve Plane Block (M-TAPA) is performed deep into the costochondral aspect at the 9th-10th costal level by injecting local anesthetics deep into the chondrium. It provides blockage of both the anterior and lateral cutaneous branches of the thoracoabdominal nerve. As there are studies showing M-TAPA block to be effective for postoperative analgesia for other abdominal surgeries, its effect on patients undergoing living liver donor surgery has not been studied yet. We hypothesize that M-TAPA block performed in living liver donors would reduce opioid consumption in the first 48 hours after surgery.

DETAILED DESCRIPTION:
Open hepatic resection for living liver transplantation donor surgery can cause severe postoperative pain and if not treated properly, may increase the risk of chronic pain development, which has a significant impact on the patient's daily life quality. The use of interfascial plane blocks for pain control has increased in recent years, as ultrasonography (USG) has become a part of daily routine. Interfascial plane blocks provide effective postoperative analgesia. Additionally, reducing postoperative opioid consumption may be a useful strategy to provide hemodynamic stability and promote early mobilization. Case reports state interfascial plane blocks to be effective and safe for providing effective analgesia compared to systemic analgesia in living liver donor surgeries. As studies are showing M-TAPA block to be effective for postoperative analgesia for other abdominal surgeries, its effect on patients undergoing living liver donor surgery has not been studied yet. We hypothesize that the M-TAPA block performed in living liver donors would reduce opioid consumption in the first 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria: Patients American Society of Anesthesiologists (ASA) classification I- II Scheduled for living liver donation surgery for liver transplantation under general anesthesia

Exclusion Criteria: Patients

* with history of bleeding diathesis,
* receiving anticoagulant treatment,
* with allergies or sensitivity to drugs used,
* with an infection on the puncture site
* who do not accept the procedure or participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Opioid consumption (Fentanyl PCA) | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, 24 and 48 hours
  The primary aim is to compare postoperative opioid consumption from the PCA device.

SECONDARY OUTCOMES:
Pain scores (Numerical rating scale-NRS | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, 24 and 48 hours]
  The secondary aim is to compare NRS at the postoperative 48 h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded.
Need for rescue analgesia (meperidine) | Postoperative 48 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 48 h.
Adverse events | Postoperative 48 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching) related to opioid use.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Mega Hospital Complex, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data(IPD)

REFERENCES:
- [Background] Yong BH, Tsui SL, Leung CC, Lo CM, Liu CL, Fan ST, Young K. Management of postoperative analgesia in living liver donors. Transplant Proc. 2000 Nov;32(7):2110. doi: 10.1016/s0041-1345(00)01592-x. No abstract available. PMID 11120091
- [Background] Hacibeyoglu G, Topal A, Arican S, Kilicaslan A, Tekin A, Uzun ST. USG guided bilateral erector spinae plane block is an effective and safe postoperative analgesia method for living donor liver transplantation. J Clin Anesth. 2018 Sep;49:36-37. doi: 10.1016/j.jclinane.2018.06.003. Epub 2018 Jun 5. No abstract available. PMID 29883965
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940
- [Background] Aikawa K, Tanaka N, Morimoto Y. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides a sufficient postoperative analgesia for laparoscopic sleeve gastrectomy. J Clin Anesth. 2020 Feb;59:44-45. doi: 10.1016/j.jclinane.2019.06.020. Epub 2019 Jun 15. No abstract available. PMID 31212124
- [Derived] Gungor H, Ince A, Ciftci B, Emre Golboyu B, Asici M, Karaaslan P, Yanaral TU. Ultrasound-Guided Modified Thoracoabdominal Nerve Block Through Perichondrial Approach for Postoperative Analgesia Management in Living Liver Donors: A Randomized, Prospective, Controlled Study. Clin Transplant. 2025 Sep;39(9):e70224. doi: 10.1111/ctr.70224. PMID 40892532